CLINICAL TRIAL: NCT00799799
Title: Adoptive Immunotherapy of High Risk Acute Myeloblastic Leukemia Patients Using Haploidentical Kir Ligand-mismatched Natural Killer Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: prof. Roberto M. Lemoli, Institute of Hematology "L. & A. Seragnoli" - University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK TRIAL
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Myeloblastic Leukemia
Keywords: Nk cells infusion; minimal residual disease in AML patients; trafficking of NK cells after infusion; cytolytic effects on leukemic cells
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NK (Experimental): patient treated as per protocol
  Interventions: Biological: NK cells

INTERVENTIONS:
Biological: NK cells — NK cells infusion after immunosuppressive chemotherapy

SUMMARY:
AML patients with de-novo or secondary disease with age greater than 18 years not eligible for stem cell transplantation for medical contraindications, lack of donor or lack of stem cells,are eligible. Leukemias other than AML and M3 FAB subtype will be excluded from the study. Immunosuppressive chemotherapy prior to NK cell infusion will include: fludarabine and cyclophosphamide 4g/m2 (Flu/Cy). The therapy will be administered over 6 days on inpatient basis. Haploidentical NK cells will be selected from a steady-state large volume leukapheresis product from a suitable KIR ligand incompatible donor. Donor-recipients pairs will be selected on the basis of known KIR ligands. In particular, haploidentical donors will be included if present at least one allele mismatch at a class I locus among the following ones: HLA-C alleles with Asn77-Lys80, HLA-C alleles with Ser77-Asn80, HLA-Bw4 alleles. Immunomagnetic enrichment of NK cells will follow two subsequent steps: 1) depletion of CD3+ T cells followed by 2) positive selection of CD56+ NK cells. Contaminating CD3+ T cells will be carefully evaluated.

DETAILED DESCRIPTION:
When previously cryproserved NK cells are still available, further re-infusions may be performed, according to PI's evaluation. The number of remaining NK cells must be sufficient for the reinfusion of at least the minimum dose of cells (106/kg). At least two months should elapse between two consecutive infusion procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Performance Status ≥ 70% (Karnofsky score) or ≤ 2 (WHO).
* Age greater than 18 years.
* Availability of a KIR incompatible haploidentical donor.
* Adequate renal (serum creatinine < 2 mg/dl), pulmonary (Sat O2 ≥ 96%) and hepatic (ALT/AST < 2.5 x N) function.
* Patients enrolled in the protocol must have an autologous graft cryopreserved to be reinfused in case of severe myelosuppression induced by haploidentical NK cells. Back-up cells will be reinfused in case of ANC < 0.5 x 109/L at day + 40 from the start of immunosuppressive regimen.

Exclusion Criteria:

* Age < 18.
* People unable to give informed consent.
* HIV positivity.
* HCV positivity with high viral load.
* Intercurrent organ damage or medical problems that would interfere with therapy.
* Pregnant or nursing females.
* Current uncontrolled infection.
* No availability of a cryopreserved autologous stem cell graft to be reinfused in case of severe myelosuppression.
* Signs or symptoms of fluid retention (e.g. pleural effusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of the selection and reinfusion of 5x10E6 haploidentical natural killer (NK) cells /Kg of body weight (target cell dose) in at least 40% of adult patients with active acute myeloblastic leukemia (AML) entering the study | every 6 months
To assess the feasibility of the reinfusion of the minimum accepted cell dose (1x10E6 haploidentical NK cells /Kg) in all patients enrolled into the protocol | every 6 months

SECONDARY OUTCOMES:
To evaluate the microchimerism of AML patients receiving haploidentical human NK cells for adoptive immunotherapy | every 6 months
To evaluate, in vitro and in vivo, the antitumor activity of haploidentical NK cells infused in AML patients | every 6 months
To assess the percentage of patients entering complete remission (CR) after the reinfusion of highly purified haploidentical NK cells | every 6 months
To assess the disease-free and overall survival of AML patients infused with haploidentical NK cells | every 6 months
To assess the safety of infusion of haploidentical NK cells, following immunosuppressive chemotherapy, considered as the incidence of adverse event (graded according to WHO) and clinically significant abnormal laboratory values following reinfusion | every 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology "L. & A. Seragnoli", Bologna, Bo, Italy

REFERENCES:
- [Background] Ruggeri L, Capanni M, Urbani E, Perruccio K, Shlomchik WD, Tosti A, Posati S, Rogaia D, Frassoni F, Aversa F, Martelli MF, Velardi A. Effectiveness of donor natural killer cell alloreactivity in mismatched hematopoietic transplants. Science. 2002 Mar 15;295(5562):2097-100. doi: 10.1126/science.1068440. PMID 11896281
- [Derived] Curti A, Ruggeri L, D'Addio A, Bontadini A, Dan E, Motta MR, Trabanelli S, Giudice V, Urbani E, Martinelli G, Paolini S, Fruet F, Isidori A, Parisi S, Bandini G, Baccarani M, Velardi A, Lemoli RM. Successful transfer of alloreactive haploidentical KIR ligand-mismatched natural killer cells after infusion in elderly high risk acute myeloid leukemia patients. Blood. 2011 Sep 22;118(12):3273-9. doi: 10.1182/blood-2011-01-329508. Epub 2011 Jul 25. PMID 21791425